CLINICAL TRIAL: NCT02831218
Title: Quantitative Coronary Angiography Versus Imaging GUIDancE for Bioresorbable Vascular Scaffold Implantation
Acronym: GUIDE-BVS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was merged into HOWTO-BRS study.
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-13
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Percutaneous Transluminal Coronary Angioplasty
Keywords: bioresorbable vascular scaffold; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- QCA and Aspirin alone (Experimental)
  Interventions: Procedure: QCA and Aspirin
- QCA and Clopidogrel alone (Experimental)
  Interventions: Procedure: QCA and Clopidogrel
- Imaging guided and Aspirin alone (Active Comparator)
  Interventions: Procedure: Imaging guided and Aspirin
- Imaging guided and Clopidogrel alone (Active Comparator)
  Interventions: Procedure: Imaging guided and Clopidogrel

INTERVENTIONS:
Procedure: QCA and Aspirin — QCA(quantitative coronary angiography) guided BVS implantation and all patients are treated with dual antiplatelet therapy (aspirin 100mg/day and clopidogrel 75mg per day[or ticagrelor 90mg po bid]) for 12 months after BVS implantation, and randomized to either aspirin alone (aspirin 100mg/day) or clopidogrel alone (clopidogrel 75mg /day) for the next 4 years.
  Arms: QCA and Aspirin alone
Procedure: QCA and Clopidogrel — QCA(quantitative coronary angiography) guided BVS implantation and all patients are treated with dual antiplatelet therapy (aspirin 100mg/day and clopidogrel 75mg per day[or ticagrelor 90mg po bid]) for 12 months after BVS implantation, and randomized to either aspirin alone (aspirin 100mg/day) or clopidogrel alone (clopidogrel 75mg /day) for the next 4 years.
  Arms: QCA and Clopidogrel alone
Procedure: Imaging guided and Aspirin — BVS size and length were selected by on-line IVUS(intravascular ultrasound) or OCT(optical coherence tomography) measurements and all patients are treated with dual antiplatelet therapy (aspirin 100mg/day and clopidogrel 75mg per day[or ticagrelor 90mg po bid]) for 12 months after BVS implantation, and randomized to either aspirin alone (aspirin 100mg/day) or clopidogrel alone (clopidogrel 75mg /day) for the next 4 years.
  Arms: Imaging guided and Aspirin alone
Procedure: Imaging guided and Clopidogrel — BVS size and length were selected by on-line IVUS(intravascular ultrasound) or OCT(optical coherence tomography) measurements and all patients are treated with dual antiplatelet therapy (aspirin 100mg/day and clopidogrel 75mg per day[or ticagrelor 90mg po bid]) for 12 months after BVS implantation, and randomized to either aspirin alone (aspirin 100mg/day) or clopidogrel alone (clopidogrel 75mg /day) for the next 4 years.
  Arms: Imaging guided and Clopidogrel alone

SUMMARY:
The purpose of this study is to compare clinical outcomes between QCA(quantitative coronary angiography)-guided and imaging-guided strategy in patients with native coronary artery disease undergoing Bioresorbable Vascular Scaffold implantation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age
* Typical chest pain or objective evidence of myocardial ischemia suitable for elective percutaneous coronary intervention
* Native coronary artery lesions with lesion length ≤ 50mm and reference vessel diameter of 2.3 - 3.75mm by QCA(quantitative coronary angiography) assessment
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Angiographic exclusion criteria: any of the followings

  1. Small vessel: mean reference size < 2.3 mm by QCA(quantitative coronary angiography)
  2. True bifurcation lesion with a large side branch (reference vessel diameter > 2.3mm) requiring a complex two-stent approach
  3. Left main lesions
  4. Ostial lesions within 3mm of the origin: right coronary artery, left anterior descending artery, or left circumflex artery
  5. Impaired delivery of the Absorb BVS is expected:
* Extreme angulation (≥90°) proximal to or within the target lesion.
* Excessive tortuosity (≥two 45° angles) proximal to or within the target lesion.
* Moderate or heavy calcification proximal to or within the target lesion. 6. In-stent restenotic lesions
* ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention (with 12- 24 hour after symptoms onset)
* Prior percutaneous coronary intervention within the target vessel during the last 12 months.
* Prior percutaneous coronary intervention within the non-target vessel or any peripheral intervention is acceptable if performed anytime >30 days before the index procedure, or between 24 hours and 30 days before the index procedure if successful and uncomplicated.
* Left ventricular ejection fraction (LVEF) < 30%
* Hypersensitivity or contraindication to device material and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated.
* Persistent thrombocytopenia (platelet count <100,000/µl)
* Any history of hemorrhagic stroke or intracranial hemorrhage, transient ischemic attack (TIA) or ischemic stroke within the past 6 months
* A known intolerance to a study drug (aspirin, clopidogrel or ticagrelor)
* Patients requiring long-term oral anticoagulants or cilostazol
* Any surgery requiring general anesthesia or discontinuation of aspirin and/or an ADP antagonist is planned within 12 months after the procedure.
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* Life expectancy < 5 years for any non-cardiac or cardiac causes
* Unwillingness or inability to comply with the procedures described in this protocol.
* Patient's pregnant or breast-feeding or child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  the cumulative incidence of cardiac death, target vessel myocardial infarction or ischemia-driven target lesion revascularization at 12 months after the index procedure.

SECONDARY OUTCOMES:
Device success | 1 day
  Successful delivery and deployment of the study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 30% by quantitative coronary angiography (QCA).
Procedural success | 24 hours
  Achievement of final in-scaffold/stent residual stenosis of less than 30% by QCA with successful delivery and deployment of at least one study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel myocardial infarction or repeat target lesion revascularization during the hospital stay (24 hour after an index procedure).
Death | 1 year and 5 years
Myocardial infarction | 1 year and 5 years
Scaffold thrombosis | 1 year and 5 years
Stroke | 1 year and 5 years
Target lesion revascularization | 1 year and 5 years
Any revascularization | 1 year and 5 years
Target lesion failure | 1 year and 5 years
  cardiac death, target vessel myocardial infarction or ischemia-driven target lesion failure
event rate of net clinical events | 5 years
  defined as composite event of cardiovascular death, myocardial infarction, stroke, clinically relevant bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.